CLINICAL TRIAL: NCT01250574
Title: Neutrophil CD64 and Procalcitonin as Novel Biomarkers for Postoperative Infections
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Tom Oresland, Professor, University Hospital, Akershus
Other Study IDs: 2010/2356
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Bacterial Infection; Postoperative Infection; Abdominal Infection
Keywords: CD64; Procalcitonin
MeSH Terms: conditions — Bacterial Infections; Intraabdominal Infections | interventions — Receptors, IgG; Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postoperative infections
  Interventions: Other: CD64 and Procalcitonin
- Bacterial infections in the GI tract
  Interventions: Other: CD64 and Procalcitonin

INTERVENTIONS:
Other: CD64 and Procalcitonin — Blood tests taken before and regularly after surgery or other treatment.
  Groups: Postoperative infections
Other: CD64 and Procalcitonin — Blood tests taken before and regularly after surgery or other treatment.
  Groups: Bacterial infections in the GI tract

SUMMARY:
Postoperative complications, especially bacterial infections, are relatively common and cause increased morbidity and mortality. Effective and timely antimicrobial treatment is important for prognosis, and delayed diagnosis and treatment substantially increase mortality. The early diagnosis of infection and sepsis are today based on diagnostic tests that have been available for years, like WBC count, SR and CRP. These markers suffer from several drawbacks; their sensitivity and specificity for infection and sepsis are not good enough and their kinetics are rather slow in terms of both increase and decrease. A major disadvantage of CRP is that after surgery and trauma this marker generally increases for several days, reaching a plateau typically on day 2-4 following the event, and therefore, in most cases do not offer the needed guidance for early treatment of bacterial infection. More recently, other biomarkers for infection and sepsis have become available, some of which appear acceptable for diagnostic use. Procalcitonin (PCT) and neutrophil CD64 are both promising new markers for the early detection of infection. They do both have their pros and cons compared to each other and compared to the traditional markers, such as CRP and WBC count. It is a general view that further research is needed before these markers will be accepted as part of the routine protocol for the diagnosis of infections, especially in relation to postoperative complications. The aim of the present study is to investigate the clinical utility of procalcitonin (PCT) and neutrophil CD64 as markers for infection and inflammation:

* to evaluate if it is possible to detect early phase postoperative infections by using these tests versus traditional markers such as CRP, SR and WBC count (with differential).
* to differentiate between systemic bacterial infection and systemic inflammation due to the surgical trauma.

The hypothesis is that PCT and neutrophil CD64 are more sensitive and specific analysis for the early detection of infection after abdominal surgery than CRP (and other widely used tests for inflammation and infection), and that neutrophil CD64 is more specific than PCT. Patients admitted to the Department of Gastroenterological Surgery, Akershus University Hospital for elective abdominal surgery will be included in the study after informed consent. Initially consecutive series of 150 patients will be included, but this number may be increased depending on the number of observed infections during the course of the study. All patients will be monitored and treated by the formal protocol related to clinical signs of infection, such as abcess, peritonitis, pneumonia, sepsis and septic shock. In addition to the analytical parameters routinely used today in order to discover infections (CRP, WBC count etc), blood samples for PCT and neutrophil CD64 will be analyzed before surgery and daily during the stay at the hospital. In the case of signs of infection, locally or systemic, the frequencies of analysing PCT and CD64 will be increased according to the severity of the changes in the clinical condition. The expression of CD64 will be measured by flow-cytometry and PCT will be measured by an immunochemical method.

ELIGIBILITY:
Inclusion Criteria:

* Suspected infection in the GI tract or after abdominal surgery

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Gastroenterological surgery
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2010-11; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Oslo, Lorenskog, Norway